CLINICAL TRIAL: NCT03095456
Title: A Phase 3b, Randomized, Double-Blind, Double-Dummy, Parallel-Group, Study to Compare Once Daily Nebulized Revefenacin With Spiriva Once Daily Delivered Via the HandiHaler® on Lung Function in Subjects With COPD and a Low PIFR
Brief Title: Revefenacin Peak Inspiratory Flow Rate (PIFR) Study in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0149
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Results first posted 2018-12-31 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD; Low Peak Inspiratory Flow Rate (PIFR)
Keywords: Chronic Obstructive Pulmonary Disease, COPD; Low Peak Inspiratory Flow Rate (PIFR)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Revefenacin (Experimental): Active Revefenacin and placebo (in place of Spiriva Handihaler®)
  Interventions: Drug: Revefenacin; Drug: Placebo for Spiriva Handihaler®
- Spiriva Handihaler® (Active Comparator): Active Spiriva Handihaler® and placebo (in place of Revefenacin)
  Interventions: Combination Product: Spiriva Handihaler®; Drug: Placebo for Revefenacin

INTERVENTIONS:
Drug: Revefenacin — Revefenacin administered via nebulization.
  Other Names: TD-4208
  Arms: Revefenacin
Combination Product: Spiriva Handihaler® — Spiriva Handihaler® contains Spiriva (also known as Tiotropium) and is administered via HandiHaler® device.
  Other Names: Tiotropium
  Arms: Spiriva Handihaler®
Drug: Placebo for Revefenacin — Placebo administered as double blind, double dummy via nebulization.
  Arms: Spiriva Handihaler®
Drug: Placebo for Spiriva Handihaler® — Placebo administered as double blind, double dummy via Spiriva HandiHaler®.
  Arms: Revefenacin

SUMMARY:
This study is a randomized, double-blind, double-dummy, parallel group study to compare once daily nebulized Revefenacin with Spiriva once daily delivered via the HandiHaler® on lung function in subjects with COPD and a Low Peak Inspiratory Flow Rate.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female subject 40 years of age or older with a diagnosis of COPD.
* Subject has a current or past cigarette smoking history (or equivalent for cigar or pipe smoking history) of at least 10 pack-years.
* Subject is willing and able to provide signed and dated written informed consent to participate prior to initiation of any study related procedures.

Exclusion Criteria:

* Subject has a concurrent disease or condition that, in the opinion of the investigator, would interfere with continued study participation or confound the evaluation of safety and tolerability of the study drug.
* Subject has a history of reactions or hypersensitivity to inhaled or nebulized anticholinergics.
* Subject suffers from any medical condition that would preclude the use of inhaled anticholinergics, including narrow-angle glaucoma, symptomatic benign prostatic hyperplasia, bladder neck obstruction, or urinary retention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-11-25 (Actual); Study Completion 2017-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Clinical Research of Rock Hill, Rock Hill, South Carolina, United States

REFERENCES:
- [Derived] Ohar JA, Mahler DA, Davis GN, Lombardi DA, Moran EJ, Crater GD. Clinical Burden of Chronic Obstructive Pulmonary Disease in Patients with Suboptimal Peak Inspiratory Flow. Can Respir J. 2024 Mar 22;2024:8034923. doi: 10.1155/2024/8034923. eCollection 2024. PMID 38560416
- [Derived] Barnes CN, Mahler DA, Ohar JA, Lombardi DA, Crater GD. Peak Inspiratory Flows: Defining Repeatability Limits and a Predictive Equation for Different Inhalers. Chest. 2020 Oct;158(4):1413-1419. doi: 10.1016/j.chest.2020.03.072. Epub 2020 Apr 25. PMID 32343967
- [Derived] Mahler DA, Ohar JA, Barnes CN, Moran EJ, Pendyala S, Crater GD. Nebulized Versus Dry Powder Long-Acting Muscarinic Antagonist Bronchodilators in Patients With COPD and Suboptimal Peak Inspiratory Flow Rate. Chronic Obstr Pulm Dis. 2019 Oct 23;6(4):321-31. doi: 10.15326/jcopdf.6.4.2019.0137. PMID 31647854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Revefenacin | Spiriva Handihaler®
Started | 103 | 104
Completed | 99 | 96
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Revefenacin | Spiriva Handihaler® | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 53 | 104
  >=65 years | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.94) | 65.1 (8.36) | 65.1 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 60 | 64 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 96 | 101 | 197
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 90 | 95 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 104 | 206
Smoking history [Count of Participants; unit: Participants]
  Current Smoker | 46 | 50 | 96
  Former Smoker | 56 | 54 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 on Day 29
Description: FEV1 = forced expiratory volume at one second
Time Frame: Baseline and Day 29
Population: Intent-to-treat (ITT) analysis set
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 89 | 90
mL | 63.0 (20.17) | 47.3 (19.06)

2. Secondary Outcome: Change From Baseline Trough FVC (Forced Vital Capacity) on Day 29
Time Frame: Baseline and Day 29
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 89 | 90
mL | 125.4 (38.75) | 55.8 (36.62)

3. Secondary Outcome: Change From Baseline Trough Inspiratory Capacity (IC) on Day 29
Time Frame: Baseline and Day 29
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 82 | 88
mL | 71.4 (42.33) | 84.1 (40.02)

4. Secondary Outcome: Change From Baseline Peak FEV1 on Day 29
Time Frame: Baseline and Day 29 (0-4 hours)
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 91 | 90
mL | 174.2 (18.70) | 197.7 (17.73)

5. Secondary Outcome: Change From Baseline Peak FVC on Day 29
Time Frame: Baseline and Day 29 (0-4 hours)
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 91 | 90
mL | 354.2 (37.35) | 340.1 (35.49)

6. Secondary Outcome: Summary of Rescue Medication Use: Puffs Per Day
Time Frame: 1 Month
Measure: Least Squares Mean (Standard Error); unit: puffs per day
Arm/Group | Revefenacin | Spiriva Handihaler®
Number analyzed (Participants) | 101 | 95
puffs per day | 3.4 (0.42) | 2.9 (0.41)

ADVERSE EVENTS:
Time Frame: From signing of ICF through the final follow-up assessment (approximately 1 month).
Arm/Group | Revefenacin | Spiriva Handihaler®
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/104
Other Adverse Events (participants affected / at risk) | 5/103 | 21/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revefenacin (N=103) | Spiriva Handihaler® (N=104)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revefenacin (N=103) | Spiriva Handihaler® (N=104)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03095456/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03095456/SAP_000.pdf